CLINICAL TRIAL: NCT03484949
Title: Randomized Trial Comparing Gastroscopy Following Web-Mediated Risk Assessment With Routine Endoscopy for Gastric Cancer Screening
Brief Title: Web-Mediated Risk Assessment for Endoscopic Screening of Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Key Laboratory of Cancer Biology (Network)
Collaborators: Tang-Du Hospital (Other); Xijing Hospital (Other)
Responsible Party: Principal Investigator, Dake Chu, Dr., Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: xjtu-20170816
Record Dates: First submitted 2018-03-25; First posted 2018-04-02 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Screening; Risk assessment
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-endoscopic screening risk assessment (Experimental)
  Interventions: Diagnostic Test: pre-endoscopic screening risk assessment
- routine screening (No Intervention)

INTERVENTIONS:
Diagnostic Test: pre-endoscopic screening risk assessment — pre-endoscopic screening risk assessment
  Arms: pre-endoscopic screening risk assessment

SUMMARY:
Gastric cancer is one of the most common malignancies in China. Early detection is critical for gastric cancer management. However, the diagnosis rate of patients with early gastric cancer is still low. Therefore, the investigator design this study to access whether pre-endoscopic screening risk assessment of genetic and environmental risk factors could improve early gastric cancer diagnosis rate.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age 18-60. 2.Signed informed consent

Exclusion Criteria:

* 1.Severe back ground disease including malignancy. 2.State after gastric surgery. 3.COPD, CHF, CRF and any disease with respiratory disturbances. 4.Deviation of the nasal septum, lack of venous access at the dorsum of the hand or any other technical problem prevents gastric acid collection or base excess evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic rate of patients with early gastric cancer | 2020
  Diagnostic rate of patients with early gastric cancer

SECONDARY OUTCOMES:
Characterization of the high-rik individual for gastric cancer | 2020
  Diagnostic rate of patients with early gastric cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Dake Chu, Xi'an, Shaanxi, China